CLINICAL TRIAL: NCT05703061
Title: Sleep in Adolescents - Pilot Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Andrea M. Spaeth, PhD, Assistant Professor, Undergraduate Academic Director, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pro2018000606
Record Dates: First submitted 2023-01-05; First posted 2023-01-27 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Sleep
MeSH Terms: interventions — Time; Beds

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to either a control group or an increased time in bed (10 hours/night) group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal Sleep Condition Group (No Intervention): This group will not partake in the intervention, they will sleep the normal amount that they do on a regular basis. Participants will wear a hip physical activity monitor and a wrist actigraph to measure sleep.
- 10-hour Time in Bed Group (Experimental): This group will partake in the intervention of increasing time in bed to 10 hours per night. Participants will wear a hip physical activity monitor and a wrist actigraph to measure sleep.
  Interventions: Behavioral: 10-hour Time in Bed

INTERVENTIONS:
Behavioral: 10-hour Time in Bed — Participants will be asked to increase their time in bed to 10-hours per night for 7 consecutive days.
  Arms: 10-hour Time in Bed Group

SUMMARY:
The goal of this pilot clinical trial is to determine the feasibility and acceptability of increasing time in bed to 10 hours per night in children aged 14-17 years. The main question it aims to answer are:

* How much additional sleep short-sleeping-adolescents (~7h TIB/night) will obtain when asked to increase time-in-bed to 10h/night for seven consecutive nights compared to those who are not asked to increase time-in-bed?
* Are adolescents able to comply with study demands: wearing two devices (one on wrist and one on hip) and completing daily sleep diaries and call-ins for seven days?
* By acquiring participant feedback, how feasible and acceptable is it to increase time in bed for sleep to 10h/night using a questionnaire and semi-structured interview?
* Complete a phone screen
* Come to Rutgers Sleep Lab for an orientation to obtain equipment, answer questionnaires and study staff will obtain consent
* Wear a wrist device and a hip device for one week to observe sleep and physical activity
* If assigned to the 10 hour time-in-bed group, they will follow specific procedures to ensure protocol adherence
* Come to the Rutgers Sleep Lab for a follow up to give back equipment and answer questionnaires

Researchers will compare the control group to the 10 hour time in bed group to see if it is feasible for 14-17 year olds to be in bed for that long and wear two devices.

DETAILED DESCRIPTION:
We are conducting this research study to determine if it is feasible to have teenagers devote more time to being in bed for sleep. Specifically, we will try to determine how much more teens sleep when spending 10 hours in bed for a week. If after it is determined from a phone screen that the child is eligible, they will be asked to come into our Center for an Orientation.

During this visit, we will explain the research study to participants and families in more detail. Families that enroll will visit the Center one more time at the end of the study. During the orientation visit, we will determine the child's final eligibility based on how much he/she sleeps and a measurement of the child's height and weight. If eligible and interested in participating, the child would wear two devices -one that measures sleep and one that measures activity - and keep a sleep diary for a week. During this week, the child would also call/text our Center twice each day to report on his/her bedtime and wake time. The second visit to the center occurs at the end of that week.

ELIGIBILITY:
Inclusion Criteria:

* Parent-reported child age of 14-17 years
* Typical sleep duration of approximately 7hr/night on school nights
* BMI for age and gender in the >5th percentile but not greater than 100% overweight.
* Parent must be the primary caretaker and at home during bed/wake times
* Reported willingness and ability to complete all study-related tasks, including wearing the wrist actigraph and hip accelerometer daily.

Exclusion Criteria:

* Diagnosable sleep disorder (including Sleep Disordered Breathing) based on parent report and participant's score on Sleep Disorders Inventory for Students-Adolescents (SDIS-A).
* Medication use or parent-reported diagnosis of a serious medical condition (including psychiatric conditions) that may impact sleep.
* Excessive intake of caffeine (>300mg/day), drug (including nicotine) or alcohol use, or a history of substance abuse.
* Actively trying to lose weight.
* Trans-meridian (east-west/west-east) travel during past month or planned travel during study time frame.
* Inability to understand or complete protocol to ensure that consent/assent and reliable and valid measures are obtained.
* Sibling of enrolled subjects, to minimize risk of bias in study findings.

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Feasibility and Acceptability of Increasing Time in Bed to 10 hours per Night in Adolescents | The questionnaire will take approximately 5-10 minutes.
  An acceptability and feasibility questionnaire will be administered to participants at a follow up visit to measure the difficulty of increasing time in bed to 10 hours per night and wearing the two devices given. This questionnaire serves as feedback for the principal investigator to measure the feasibility of adolescents increasing time in bed to 10 hours per night and wearing two devices. Roughly half the questions are open ended and gauge the participants' physical experience during the study. The other half are scored 0-4 and ask about the participants' increase or decrease in school performance, overall mental health status, and physical health status during the day. For the questions that rank 0-4, a 0 indicates that specific aspect became a lot worse since the study, and a 4 indicates it became a lot better, or it increased over the course of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Spaeth, Ph.D, Principal Investigator — Associate Professor, Lab Director
Locations (1):
- Rutgers Sleep Lab, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data that will be collected will be shared with other researchers, after deidentification.
Supporting Information: Study Protocol, ICF
Time Frame: Immediately following publication.
Access Criteria: Anyone who wishes to access the data can do so.

REFERENCES:
- [Background] Luginbuehl M B-KK, Ferron J, Anderson WM, Benbadis SR. Pediatric sleep disorders: Validation of the SleepDisorders Inventory for Students. . School Psychol Rev. 2008; 37(3):409-31.
- [Background] Actigraph Data Collection, Proofing, and Scoring Procedures AW2 2018
- [Background] Santos-Lozano A, Santin-Medeiros F, Cardon G, Torres-Luque G, Bailon R, Bergmeir C, Ruiz JR, Lucia A, Garatachea N. Actigraph GT3X: validation and determination of physical activity intensity cut points. Int J Sports Med. 2013 Nov;34(11):975-82. doi: 10.1055/s-0033-1337945. Epub 2013 May 22. PMID 23700330
- See also: Sleep Disorders Inventory for Students — https://www.sleepinventory.com/

DOCUMENTS (1):
  • Study Protocol (2022-11-04): https://cdn.clinicaltrials.gov/large-docs/61/NCT05703061/Prot_000.pdf